CLINICAL TRIAL: NCT00739362
Title: The Effects of Transcranial Direct Current Stimulation (TDCS) on Food Intake and Weight Loss
Brief Title: Effects of Brain Stimulation on Food Intake and Behavioral Weight Loss Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 999908191; 08-DK-N191
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-23

CONDITIONS: Electric Stimulation Therapy; Obesity; Weight Loss; Eating
Keywords: Behavioral Weight Loss Treatment; Obesity; Appetite Control; Weight Loss; Transcranial Direct Current Stimulation (TDCS)
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1-Sham (Sham Comparator): Active tDCS stimulation
  Interventions: Device: Transcranial Direct Current Stimulation (TDCS)
- 2-Active (Active Comparator): Active tDCS stimulation
  Interventions: Device: Transcranial Direct Current Stimulation (TDCS)
- 2-Sham (Sham Comparator): Sham/no-stimulation
  Interventions: Other: Sham/no-stimulation
- 3-Active (Active Comparator): Active tDCS stimulation
  Interventions: Device: Transcranial Direct Current Stimulation (TDCS)
- 3-Sham (Sham Comparator): Sham/no-stimulation
  Interventions: Other: Sham/no-stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (TDCS) — Active tDCS (anodal left DLPFC)
  Arms: 1-Sham; 2-Active; 3-Active
Other: Sham/no-stimulation — Sham tDCS
  Arms: 2-Sham; 3-Sham

SUMMARY:
This study will determine whether electrical stimulation of an area of the brain called the dorsolateral prefrontal cortex, which is important in determining the feeling of fullness after eating, affects how much food a person eats and weight loss over 4 weeks. It will also compare weight changes in people who attend weight loss counseling sessions and those who do not over this period of time.

Obese, non-diabetic people between 18 and 60 years of age who are in good health and who live in the Phoenix, AZ, metropolitan area are eligible for this study. Candidates must have a body mass index of 35 kg/m(2) or more and weigh less than 350 pounds.

Participants are admitted to the NIH inpatient unit in Phoenix for the first 9 days of the study for tests, which include meal tests to determine eating behaviors and caloric intake, blood and urine tests, glucose tolerance test, weight measurement, psychological assessments and DEXA scan to measure body fat. For 3 of the days, they will be asked to eat all of their food from automated vending machines. Some subjects receive transcranial direct current stimulation (TDCS). For this procedure, electrodes that conduct electricity are placed on the head and arm and the current is turned on for 40 minutes. Some tingling may be felt under the electrodes. Other subjects receive sham TDCS, with the current turned on only very briefly.

After the evaluations, subjects are discharged home from the NIH unit and instructed to eat 25 percent fewer calories than they consumed while on a weight maintenance diet the first 3 days of their inpatient stay. They maintain the lower calorie diet at home for 4 weeks. During this period they come to the NIH unit 3 days a week to receive either real or sham TDCS.

...

DETAILED DESCRIPTION:
In our studies of brain function examining areas related to hunger and fullness, a part of the brain called the left dorsolateral prefrontal cortex (DLPFC) was found to be less active in obese versus lean individuals following a meal. Furthermore, in women who have lost and maintained weight loss, the activity in this area following a meal is similar to that of lean women, suggesting that the activity in this area may improve with weight loss. Two recent studies have demonstrated a lack of increase in food craving following non-invasive brain stimulation to the left DLPFC when compared to a sham control group that did not receive brain stimulation.

The aim of our protocol is to investigate the effectiveness of one type of noninvasive brain stimulation technique, transcranial direct current stimulation (tDCS) on food intake in significantly overweight (BMI >= 30 kg/m^2) individuals. In study 1, we enrolled individuals who previously participated in this study and examined how anodal (active) stimulation or sham (no stimulation) to the left DLPFC compared to their previous stimulation condition in terms of both weight loss and food intake. The aim of Study 2 was to compare active versus sham anodal left DLPFC stimulation in a new group of volunteers.

Study 3 will be a 9-week double-blind parallel outpatient study where volunteers will come to the Clinical Research Unit 3x per week and be randomized to receive either active tDCS or "no stimulation" (sham) to the left DLPFC for stimulation sessions while being asked to follow diet that is a 25% reduction from their calculated weight maintenance calories. The primary outcome measurement will be total food (kcal) intake during a snack food taste test and weight change. Volunteers will also undergo 4 sessions of brain imaging (called functional MRI) to help us understand how the stimulation is working. Participants will also be asked to come back to the Unit after 6 months and 1 year for weight measurements. We will also examine appetitive hormones, neurocognitive and behavioral factors, which might also mediate potential changes in food intake and weight following tDCS to the left DLPFC. Positive findings from this study could demonstrate the utility of a novel and safe treatment for severe obesity. Future studies could include longer clinical trials of tDCS with extended follow-up durations.

ELIGIBILITY:
* INCLUSION CRITERIA:
* BMI >= 25 kg/m^2
* Age 18-60 years. Women who are post-menopausal will be excluded from the study due to changes in their metabolism that could affect weight loss. We will set the cutoff at age 60 so that the age difference between the men and women is not too great for analysis purposes. Minors under the age of 18 will be excluded because the time requirements of the study are such that they would interfere with school schedules.
* Right-handedness (because the treatment will be given to the left dorsolateral prefrontal cortex and the evidence accumulated in this region was only in right-handed individuals).
* Weight stable (+/- 5 percent) for last 3 months as determined by volunteer report.

EXCLUSION CRITERIA:

* Weight > 300 lbs (136 kg), as this is the general size limit of the fMRI machine. Participants >300 pounds may be included if their body habitus will allow them to fit within the diameter of the MRI machine. This will be determined on a case-by-case basis after consultation with staff at Banner Health Neuroimaging Center.
* Use of medication affecting metabolism and appetite in the last three months
* Current pregnancy, pregnancy within the past 6 months or currently lactating
* History or clinical manifestations of acute or chronic disorders or conditions that may affect appetite or energy expenditure (such as, but not limited to type 1 or type 2 diabetes, Cushing s disease, thyroid disorders, coccidiomycoses)
* Gastrointestinal disease, including inflammatory bowel diseases (e.g. Chron s disease and ulcerative colitis), malabsorption syndromes (e.g. celiac disease), gastric ulcer (active) which may alter metabolism
* Current, unstable medical conditions such as hepatitis, renal insufficiency, cancer requiring treatment in the last 5 years, or central nervous system disorders etc. as assessed by history and physical exam
* Evidence of alcohol abuse as defined by >= 8 point score on the Alcohol consumption screening AUDIT questionnaire in adults
* Evidence of drug use such as amphetamines, cocaine, heroin, or marijuana
* Current use of tobacco products that exceed "Very Low Dependence" on the Fagerstr(SqrRoot)(Delta)m Test for Nicotine Dependence Tool (score greater than 2)
* Postmenopausal women or symptoms of perimenopause (e.g. hot flashes, onset of irregular periods following age 40, elevation of FSH >20 IU following age 40 years)
* Any conditions contraindicated for MRI (e.g., pacemaker, metal in the cranial cavity, significant claustrophobia, holes in the skull made by trauma or surgery)
* Any condition not specifically mentioned above that, in the opinion of the investigator, may interfere with the study or prove unsafe for participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Estimated)
Dates: Start 2009-01-19 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
weight loss | Baseline, week 9
  Weight (kg)
food intake | Baseline, week 9
  Total energy intake during snack food taste test
brain fMRI activation in the left DLPFC when shown food vs. nonfood visual cues | Weeks 1 and 9
  Percent signal change in the left DLPFC when shown food vs. nonfood visual cues

SECONDARY OUTCOMES:
weight loss | Baseline, 6 months
  weight (kg)
responses to Iowa Gambling Task | Percent signal change in the left DLPFC when shown food vs. nonfood visual cues, appetitive hormone levels measured in blood
  Percent signal change in the left DLPFC when shown food vs. nonfood visual cues, performance on questionnaires
responses to Three Factor Eating Questionnaire | Baseline, week 9
  Percent signal change in the left DLPFC when shown food vs. nonfood visual cues, performance on questionnaires
responses to MacArthur Scale of Subjective Social Status | Baseline, week 9
  Percent signal change in the left DLPFC when shown food vs. nonfood visual cues, performance on questionnaires
responses to Gormally Binge Eating Questionnaire | Baseline, week 9
  Percent signal change in the left DLPFC when shown food vs. nonfood visual cues, performance on questionnaires
weight loss | Baseline, 1 year
  weight (kg)
responses to Perceived Stress Scale | Baseline, week 9
  Percent signal change in the left DLPFC when shown food vs. nonfood visual cues, performance on questionnaires
GLP-1 | Weeks 1 and 9
  Percent signal change in the left DLPFC when shown food vs. nonfood visual cues, appetitive hormone levels measured in blood
responses to Go/No Go Task | Percent signal change in the left DLPFC when shown food vs. nonfood visual cues, appetitive hormone levels measured in blood
  Percent signal change in the left DLPFC when shown food vs. nonfood visual cues, performance on questionnaires
Ghrelin | Weeks 1 and 9
  Percent signal change in the left DLPFC when shown food vs. nonfood visual cues, appetitive hormone levels measured in blood
macronutrient preferences | Baseline, week 9
  Percent signal change in the left DLPFC when shown food vs. nonfood visual cues, macronutrient preferences determined during snack food taste test

CONTACTS AND LOCATIONS:
Overall Officials: Marci E Gluck, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gluck ME, Alonso-Alonso M, Piaggi P, Weise CM, Jumpertz-von Schwartzenberg R, Reinhardt M, Wassermann EM, Venti CA, Votruba SB, Krakoff J. Neuromodulation targeted to the prefrontal cortex induces changes in energy intake and weight loss in obesity. Obesity (Silver Spring). 2015 Nov;23(11):2149-56. doi: 10.1002/oby.21313. PMID 26530931
- [Background] Le DS, Pannacciulli N, Chen K, Salbe AD, Del Parigi A, Hill JO, Wing RR, Reiman EM, Krakoff J. Less activation in the left dorsolateral prefrontal cortex in the reanalysis of the response to a meal in obese than in lean women and its association with successful weight loss. Am J Clin Nutr. 2007 Sep;86(3):573-9. doi: 10.1093/ajcn/86.3.573. PMID 17823419
- [Background] Heinitz S, Reinhardt M, Piaggi P, Weise CM, Diaz E, Stinson EJ, Venti C, Votruba SB, Wassermann EM, Alonso-Alonso M, Krakoff J, Gluck ME. Neuromodulation directed at the prefrontal cortex of subjects with obesity reduces snack food intake and hunger in a randomized trial. Am J Clin Nutr. 2017 Dec;106(6):1347-1357. doi: 10.3945/ajcn.117.158089. Epub 2017 Oct 18. PMID 29046305
- [Derived] Stinson EJ, Travis KT, Magerowski G, Alonso-Alonso M, Krakoff J, Gluck ME. Improved food Go/No-Go scores after transcranial direct current stimulation (tDCS) to prefrontal cortex in a randomized trial. Obesity (Silver Spring). 2022 Oct;30(10):2005-2013. doi: 10.1002/oby.23529. Epub 2022 Sep 2. PMID 36052819